CLINICAL TRIAL: NCT05740150
Title: The Efficacy of a Lock Solution Containing Taurolidine, Citrate and Heparin for the Prevention of Tunneled Central Line-associated Bloodstream Infections in Pediatric Oncology Patients, a Randomized Controlled, Mono-center Trial.
Brief Title: Central Line-associated Bloodstream Infection Prevention Using TauroLock-Hep100 in Pediatric Oncology Patients.
Acronym: CATERPILLAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: Dutch Cancer Society (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL2365.041.26; NTR668 (Registry Identifier: Nederlands Trial Register); 12617 (Other Grant/Funding Number: Dutch Cancer Society)
Record Dates: First submitted 2023-02-02; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI)
Keywords: Central Line-associated Bloodstream Infection; Paediatric oncology patients; Central venous access device
MeSH Terms: interventions — Vascular Access Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TauroLock-Hep100 (taurolidine 1.35%, citrate 4%, heparin 100 IU/mL) (Experimental)
  Interventions: Device: TauroLock-Hep100 (taurolidine 1.35%, citrate 4%, heparin 100 IU/mL)
- Heparin lock (heparin 100 IU/mL) (Active Comparator)
  Interventions: Device: Heparin lock (heparin 100 IU/mL)

INTERVENTIONS:
Device: TauroLock-Hep100 (taurolidine 1.35%, citrate 4%, heparin 100 IU/mL) — The TauroLock-Hep100 is a lock solution that is instilled in the lumen of a central venous access device after a treatment cycle.
  Arms: TauroLock-Hep100 (taurolidine 1.35%, citrate 4%, heparin 100 IU/mL)
Device: Heparin lock (heparin 100 IU/mL) — The Heparin lock is a lock solution that is instilled in the lumen of a central venous access device after a treatment cycle.
  Arms: Heparin lock (heparin 100 IU/mL)

SUMMARY:
The goal of this assessor blinded randomized controlled trial is to compare a lock solution containing taurolidine, citrate and heparin to a heparin only lock solution for the prevention of central line associated bloodstream infections in paediatric oncology patients with a central venous access device.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 - <19 years
* Radiological, cytological or histological proven paediatric malignancy (hematologic, solid, and neurologic malignancies)
* Tunnelled external central venous access device or totally implantable venous access port to be inserted at the Princess Máxima Center for Pediatric Oncology
* Planned central venous access device insertion of >90 days
* Written consent signed according to local law and regulations
* Parents/guardians or patient are willing and able to comply with the trial procedure

Exclusion Criteria:

* A previous central venous access device removed < 12 months ago.
* Expected treatment for a majority of the follow-up time in a different hospital than the Princess Maxima Center for pediatric oncology in the first 90 days of inclusion resulting in difficulties/the inability to visit the Princess Maxima Center at least once every 3 weeks.
* Primary immunological disorder
* Contra indications: known hypersensitivity to taurolidine, citrate or heparin, and a history of heparin-induced thrombocytopenia.
* Documented bacteremia in the period from 24h before catheter insertion until inclusion

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 462 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of central line associated bloodstream infections | From central venous access device insertion until the end of follow-up (maximum of 90 days).

SECONDARY OUTCOMES:
Time to first central line associated bloodstream infection | From central venous access device insertion until the end of follow-up (maximum of 90 days).
Central line associated bloodstream infection incidence per 1,000 central venous access device-days | From central venous access device insertion until the end of follow-up (maximum of 90 days).
Incidence of symptomatic central venous thrombosis | From central venous access device insertion until the end of follow-up (maximum of 90 days).
Incidence of bacteraemia | From central venous access device insertion until the end of follow-up (maximum of 90 days).
Incidence of local infections | From central venous access device insertion until the end of follow-up (maximum of 90 days).
Dispense of thrombolysis/systemic antibiotic treatment due to central line associated bloodstream infections/ central venous thrombosis | From central venous access device insertion until the end of follow-up (maximum of 90 days).
Incidence of and reasons for central venous access device-removal | From central venous access device insertion until the end of follow-up (maximum of 90 days).
Cultured microorganisms causing central line associated bloodstream infections | From central venous access device insertion until the end of follow-up (maximum of 90 days).
Days of hospital admission due to central line associated bloodstream infections/ central venous thrombosis | From central venous access device insertion until the end of follow-up (maximum of 90 days).
Safety in terms of known side effects, severe adverse events, intensive care unit admission, and mortality rate due to central line associated bloodstream infections/central venous thrombosis | From central venous access device insertion until the end of follow-up (maximum of 90 days).

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Máxima Center for Pediatric Oncology, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The results of this trial will be published in an open access peer-reviewed journal, presented at international congresses and subsequently the data (stored for at least 15 years) will be made available after publication of the main results manuscript upon reasonable requests. The patient society (Vereniging Kinderkanker Nederland) will be involved in the plan for the dissemination of the trial results to the participants and public after completion of the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before the end of the study the study protocol, statistical analysis plan and informed consent forms will be published in a peer-reviewed journal. The results of this trial will be published in an open access peer-reviewed journal, presented at international congresses and subsequently the data (stored for at least 15 years) will be made available after publication of the main results manuscript upon reasonable requests. The patient society (Vereniging Kinderkanker Nederland) will be involved in the plan for the dissemination of the trial results to the participants and public after completion of the trial.

REFERENCES:
- [Derived] van den Bosch CH, Loeffen Y, van der Steeg AFW, van der Bruggen JT, Frakking FNJ, Fiocco M, van de Ven CP, Wijnen MHWA, van de Wetering MD. CATERPILLAR-study protocol: an assessor-blinded randomised controlled trial comparing taurolidine-citrate-heparin to heparin-only lock solutions for the prevention of central line-associated bloodstream infections in paediatric oncology patients. BMJ Open. 2023 Mar 21;13(3):e069760. doi: 10.1136/bmjopen-2022-069760. PMID 36944461